CLINICAL TRIAL: NCT05549310
Title: Long-term Effect of High Flow Nasal Canula Therapy on Obstructive Sleep Apnea
Acronym: HFNC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022037
Record Dates: First submitted 2022-08-14; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-07

CONDITIONS: Obstructive Sleep Apnea; High Flow Nasal Canula; Continuous Positive Airway Pressure Ventilation
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Subjects are divided into 2 groups:HFNC group and CPAP group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP group (Active Comparator): CPAP group : The first stage:receiving CPAP treatment for 6 hours / night, for 1 month. Patients in the treatment group first use pressure titration, select the appropriate pressure after treatment.
  The second stage ( cohort study ) : After one month of the first stage of treatment, patients voluntarily continued to receive treatment and observers were included in the second stage of treatment. CPAP group continued to receive corresponding treatment for 6 months.
  Interventions: Device: CPAP
- HFNC group (Experimental): HFNC group : The first stage:receiving HFNC treatment for 6 hours / night, for 1 month. Patients in the treatment group first use pressure titration, select the appropriate pressure after treatment.
  The second stage ( cohort study ) : After one month of the first stage of treatment, patients voluntarily continued to receive treatment and observers were included in the second stage of treatment. HFNC group continued to receive corresponding treatment for 6 months.
  Interventions: Device: high-flow nasal canula oxygen therapy

INTERVENTIONS:
Device: CPAP — At the beginning of the experiment we will choose the most suitable pressure and flow for the patient by titration，
  Arms: CPAP group
Device: high-flow nasal canula oxygen therapy — At the beginning of the experiment we will choose the most suitable pressure and flow for the patient by titration，
  Arms: HFNC group

SUMMARY:
Patients meeting the criteria of obstructive sleep apnea were included, and all patients signed informed consent, which met the requirements of the ethics Committee of our unit. All subjects were hospitalized patients. Subjects were randomly enrolled into High-flow Nasal Cannula Oxygen Therapy group or Continuos Positive Airway Pressure group for 1 month of treatment. Sleep respiration monitoring data including AHI, blood oxygen saturation decline index (ODI) and minimum blood oxygen saturation were recorded before and after treatment.

After one month of the first stage of treatment, patients voluntarily continued to receive treatment and observers were included in the second stage of treatment. HFNC group and CPAP group continue to receive corresponding treatment for 6 months.Before and after the study, sleep respiratory monitoring datas,treatment failure rate，good compliance rate are recorded.

DETAILED DESCRIPTION:
Patients meeting the criteria of obstructive sleep apnea were included, and all patients signed informed consent, which met the requirements of the ethics Committee of our unit. All subjects were hospitalized patients. Subjects were randomly enrolled into High-flow Nasal Cannula Oxygen Therapy group or Continuos Positive Airway Pressure group.

Procedure

1. The first stage ( RCT study ) : subjects were divided into HFNC group and CPAP group, HFNC group received HFNC treatment 6 hours / night, 1 month ; CPAP group : receiving CPAP treatment for 6 hours / night, for 1 month. Patients in the treatment group first use pressure titration, select the appropriate pressure after treatment.

   Patients receiving CPAP treatment were enrolled in the study. Pressure titration was used first, and appropriate pressure was selected before treatment. The initial gas flow rate of patients receiving HFNC treatment was set to 30 - 40 L / min, and FiO2 was titrated to maintain the pulse oxygen saturation above 92 %, which was adjusted according to the patient 's tolerance and comfort.Record nightly sleep respiratory monitoring data, including 1 sleep characteristics : total sleep time, REM time, NREM time, sleep efficiency ( SE ) ; 2 awakening time, awakening index ( Arl ) ; aHI, average apnea time, longest apnea time ; 4 the cumulative time of average oxygen saturation, minimum oxygen saturation, ODI, and oxygen saturation below 90 % ; 5 heart rate, blood pressure, etc.
2. The second stage ( cohort study ) : After one month of the first stage of treatment, patients voluntarily continued to receive treatment and observers were included in the second stage of treatment. HFNC group and CPAP group continued to receive corresponding treatment for 6 months. Follow-up after each stage of treatment, recording sleep respiratory monitoring data, including the main endpoint : 1 Treatment failure rate 2.treatment compliance

ELIGIBILITY:
Inclusion Criteria:

meet any one of these

* There were typical symptoms of sleep snoring at night with apnea and daytime sleepiness (ESS score ≥9). Stenosis and obstruction in any part of the upper airway were observed on physical examination, with AHI≥5 times /h.

  * For patients with no significant daytime sleepiness (ESS score < 9), AHI≥10 times /h; ③ Patients with AHI≥5 times /h had one or more OSAHS complications, such as cognitive impairment, hypertension, coronary heart disease, cerebrovascular disease, diabetes and insomnia.

Exclusion Criteria:

meet any one of these

1. Patients who cannot tolerate non-invasive ventilator or transnasal high-flow oxygen therapy.
2. Ongoing treatment may affect sleep, such as sedatives, hypnotics, muscle relaxants, etc.
3. Hemodynamic instability;
4. Severe respiratory diseases;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
AHI | Change from Baseline AHI data at 1 month and 6 months.
  The data of the patient's AHI will be collected to evaluate the change of the patient's sleep.
Treatment failure rate | about sixth month
  The data of the patient's AHI will be collected to evaluate the change of the patient's device adaptation.
Good compliance rate | about sixth month
  refers to the replacement of patients during treatment to another group of respiratory support or patients give up treatment
mean apnea time | Change from Baseline mean apnea time data at 1 month and 6 months.
  The data of the patient's mean apnea time will be collected to evaluate the change of the patient's sleep.
longest apnea time | Change from Baseline longest apnea time data at 1 month and 6 months.
  The data of the patient's mean apnea time will be collected to evaluate the change of the patient's sleep.
Mean oxygen saturation | Change from Baseline Mean oxygen saturation data at 1 month and 6 months.
  The data of the patient's mean apnea time will be collected to evaluate the change of the patient's oxygen saturation.
minimum oxygen saturation | Change from Baseline minimum oxygen saturation data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's oxygen saturation.
ODI | Change from Baseline ODI data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's oxygen saturation.
oxygen saturation < 90 % cumulative timesaturation | Change from Baseline oxygen saturation < 90 % cumulative timesaturation data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's oxygen saturation.
Gender | by experiment finished:about 1 year
  general condition
age | by experiment finished:about 1 year
  general condition
height | by experiment finished:about 1 year
  general condition
weight | by experiment finished:about 1 year
  general condition

SECONDARY OUTCOMES:
total sleep time | Change from Baseline total sleep time data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's sleep.
REM time | Change from Baseline REM time data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's sleep.
NREM time | Change from Baseline NREM time data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's sleep.
sleep efficiency ( SE ) | Change from Baseline sleep efficiency ( SE ) data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's sleep.
awakening time | Change from Baseline awakening time data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's sleep.
awakening index ( Arl ) | Change from Baseline awakening index ( Arl ) data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's sleep.
heart rate | Change from Baseline heart rate data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's circulation condition.
blood pressure | Change from Baseline blood pressure data at 1 month and 6 months.
  The data will be collected to evaluate the change of the patient's circulation condition..

CONTACTS AND LOCATIONS:
Overall Officials: Zhuo Han, master, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jordan AS, McSharry DG, Malhotra A. Adult obstructive sleep apnoea. Lancet. 2014 Feb 22;383(9918):736-47. doi: 10.1016/S0140-6736(13)60734-5. Epub 2013 Aug 2. PMID 23910433
- [Background] Benjafield AV, Ayas NT, Eastwood PR, Heinzer R, Ip MSM, Morrell MJ, Nunez CM, Patel SR, Penzel T, Pepin JL, Peppard PE, Sinha S, Tufik S, Valentine K, Malhotra A. Estimation of the global prevalence and burden of obstructive sleep apnoea: a literature-based analysis. Lancet Respir Med. 2019 Aug;7(8):687-698. doi: 10.1016/S2213-2600(19)30198-5. Epub 2019 Jul 9. PMID 31300334
- [Background] Parke RL, McGuinness SP. Pressures delivered by nasal high flow oxygen during all phases of the respiratory cycle. Respir Care. 2013 Oct;58(10):1621-4. doi: 10.4187/respcare.02358. Epub 2013 Mar 19. PMID 23513246
- [Background] Nakanishi N, Suzuki Y, Ishihara M, Ueno Y, Tane N, Tsunano Y, Itagaki T, Oto J. Effect of High-Flow Nasal Cannula on Sleep-disordered Breathing and Sleep Quality in Patients With Acute Stroke. Cureus. 2020 Jul 20;12(7):e9303. doi: 10.7759/cureus.9303. PMID 32832300
- [Background] Nilius G, Wessendorf T, Maurer J, Stoohs R, Patil SP, Schubert N, Schneider H. Predictors for treating obstructive sleep apnea with an open nasal cannula system (transnasal insufflation). Chest. 2010 Mar;137(3):521-8. doi: 10.1378/chest.09-0357. Epub 2009 Dec 1. PMID 19952061
- [Result] Yan H, Qinghua L, Mengyuan P, Yaoyu C, Long Z, Mengjie L, Xiaosong D, Fang H. High flow nasal cannula therapy for obstructive sleep apnea in adults. Sleep Breath. 2022 Jun;26(2):783-791. doi: 10.1007/s11325-021-02453-6. Epub 2021 Aug 12. PMID 34383275